CLINICAL TRIAL: NCT02927444
Title: Multi-Center, Randomized, Double-Blind, Phase III Trial to Assess the Immunogenicity and Safety of Booster Vaccination With NBP606 in Healthy Toddlers (The Extension Study of NBP606_PCVI_III_2013)
Brief Title: Immunogenicity and Safety Study of NBP606 in Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NBP606_PCVT_III_2013
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2017-10

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NBP606 (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: NBP606
- Prevnar13 (Active Comparator): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: Prevnar13

INTERVENTIONS:
Biological: NBP606 — A single intramuscular injection into the thigh
  Arms: NBP606
Biological: Prevnar13 — A single intramuscular injection into the thigh
  Arms: Prevnar13

SUMMARY:
This study will assess the immunogenicity and safety of booster vaccination with NBP606 compared to the existing commercial vaccine, when given concomitantly with routine pediatric vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants who completed 3 doses of primary vaccination (NBP606_PCVI_III_2013), available for follow-ups during the study period.
* The LAR (Legally Authorized Representative) who understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

* Administration of other vaccines, except the ones provided in this study, within 1month prior to booster study
* Known hypersensitivity to any components of the pneumococcal vaccine
* Any confirmed or suspected immunosuppressive or immunodeficient conditions
* Coagulation disorder contraindicating IM(intramuscular) vaccination
* Participation to another study

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 462 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with the targeted antibody concentration | 1 month after the booster vaccination

SECONDARY OUTCOMES:
Geometric mean concentration ratio | 1 month after the booster vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Seoul, South Korea